CLINICAL TRIAL: NCT05779683
Title: Validation Of Cardiac Output Using Pulse Decomposition Analysis In Post-Cardiac Surgery Patients In The ICU
Brief Title: Caretaker in the Cardiovascular Intensive Care Unit (CVICU)
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00074289
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Output; Hemodynamic Monitoring
Keywords: cardiopulmonary bypass; Blood Pressure (BP) monitoring; Pulmonary Artery (PA) catheters

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Caretaker device in CVICU patient: device placed on the subject after arrival to the cardiac intensive care unit postoperatively
  Interventions: Device: Caretaker Device placement

INTERVENTIONS:
Device: Caretaker Device placement — placement of the device on the postoperative cardiac surgery patient that has a pulmonary artery catheter for comparison readings

SUMMARY:
To monitor the cardiac post-op patient population with both the pulmonary artery catheter (PAC) and the Caretaker monitor, which will seek to validate the Caretaker monitor against continuous CO via the PAC. Up to a third of post-operative cardiac surgery patients develop cardiac arrhythmias such as atrial flutter and atrial fibrillation. Secondary analysis will be performed on the collected data to assess the Caretaker monitor's agreement with the PAC during periods of arrhythmia. Successful completion this study will provide clinical validation of the Caretaker monitor in one of the most hemodynamically challenging patient populations (post-cardiac surgery patients in the ICU), including during arrhythmias. The Caretaker monitor is most beneficial as it is non-invasive, is a minimal risk device, and for this protocol will not be utilized to make treatment decisions for the study subject. This device also does not project energy into the subject.

DETAILED DESCRIPTION:
Up to a third of post-operative cardiac surgery patients develop cardiac arrhythmias such as atrial flutter and atrial fibrillation. Secondary analysis will be performed on the collected data to assess the Caretaker monitor's agreement with the PAC during periods of arrhythmia. Successful completion this study will provide clinical validation of the Caretaker monitor in one of the most hemodynamically challenging patient populations (post-cardiac surgery patients in the ICU), including during arrhythmias. The Caretaker monitor is most beneficial as it is non-invasive, is a minimal risk device, and for this protocol will not be utilized to make treatment decisions for the study subject. This device also does not project energy into the subject.

ELIGIBILITY:
Inclusion:

* Adult post-cardiac surgery needing cardiopulmonary bypass and use of the PAC as standard of care, (s/p Coronary artery bypass graft surgery (CABG), valve, heart transplant, major aortic & other vascular surgery, and a combination of CABG and valve procedures)
* patients (age > 18) admitted to the Intensive Care Unit (ICU)
* Pulmonary artery catheter (continuous or intermittent thermodilution cardiac output) and an arterial catheter for Blood Pressure monitoring (standard of care)

Exclusion:

* Patients without an appropriately positioned or functioning PA catheter admitted to the cardiac surgery ICU after surgery
* Patients on left ventricular assist device (LVAD) support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult post-cardiac surgery needing cardiopulmonary bypass and use of the PAC as standard of care, (s/p CABG, valve, heart transplant, major aortic & other vascular surgery, and a combination of CABG and valve procedures)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Comparison of hemodynamic readings between the Caretaker and the PAC | 24 hours
  To assess the agreement of the Caretaker monitor CO with the thermodilution method using the swan-ganz or pulmonary artery (PAC) catheter in critically ill cardiac surgery post-op ICU patients.
Number of Periods of Carbon monoxide (CO) Instability | 24 hours
  The incidence of CO instability after removal of PAC. Comparison of hemodynamic readings after removal of the PAC between the Caretaker and vital signs obtained as standard of care
Time Spent in Periods of CO Instability | 24 hours
  The time spent during periods of CO instability after removal of PAC. Comparison of hemodynamic readings after removal of the PAC between the Caretaker and vital signs obtained as standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Khanna, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT05779683/ICF_000.pdf